CLINICAL TRIAL: NCT00941096
Title: Efficacy Of The Bimatoprost/Timolol Fixed Combination In Patients Treated With Bimatoprost for Primary Open Angle Glaucoma, Exfoliation Glaucoma or Ocular Hypertension.
Brief Title: Intraocular Pressure Reduction With the Bimatoprost/Timolol Fixed Combination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Responsible Party: Andreas Katsanos, MD, PhD, Larissa University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 17062009-136
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular Hypertension; Lumigan; Ganfort
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Bimatoprost; Ganfort

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Drug: Bimatoprost and Bimatoprost/Timolol fixed combination. — Following an appropriate wash-out period, participants were given a 5-week long treatment with Bimatoprost 0.03% once daily in the evening followed by a further 5-week long treatment with the Bimatoprost 0.03%/Timolol 0.5% fixed combination administered in the evening.
  Other Names: Lumigan; Ganfort

SUMMARY:
The purpose of this study is to examine the ocular hypotensive effect of Bimatoprost and the potential additional effect of the Bimatoprost/Timolol fixed combination in eyes with ocular hypertension, primary open angle glaucoma or exfoliation glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma
* Exfoliation glaucoma
* Ocular hypertension

Exclusion Criteria:

* Younger than 18 years old
* Inability to understand and/or follow study requirements
* Women of childbearing potential not using reliable birth control, pregnant or lactating women
* History of chronic obstructive pulmonary disease, heart failure, 2nd or 3rd AV block
* Anticipated modification of treatment for systemic hypertension during the study period
* History of ocular herpes, corneal scarring, conventional or laser surgery or macular pathology
* History of allergy, poor tolerability or poor response to study medication
* Best corrected visual acuity less than 0.4
* Significant visual field defect (MD<15.0 dB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Mean diurnal intraocular pressure | Five weeks on each medication

CONTACTS AND LOCATIONS:
Locations (1):
- University Eye Clinic, Larissa, Thessaly, Greece